CLINICAL TRIAL: NCT03132584
Title: Ph1 Cyclophosphamide & Alemtuzumab in CD52+ R/R Double-Hit, Diffuse Lg B-cell or High Gr B-cell Lymphomas, NOS With MYC & BCL2 Over-expression, MYC-Positive Transformed Follicular Lymphoma, & CD52+ Mature T-cell Lymphoproliferative Disorder
Brief Title: Cyclophosphamide and Alemtuzumab In Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Genzyme, a Sanofi Company (Industry); Sanofi (Industry)
Responsible Party: Principal Investigator, Ann S. LaCasce, MD, Prinicipal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-034
Record Dates: First submitted 2017-04-24; First posted 2017-04-28 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Non Hodgkin Lymphoma; High-grade B-cell Lymphoma; Diffuse Large B Cell Lymphoma
Keywords: Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse | interventions — Cyclophosphamide; Alemtuzumab

STUDY DESIGN:
Intervention Model Description: This is a phase I study in the standard 3+3 dose escalation design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cyclophosphamide and Alemtuzumab (Experimental): After the screening procedures confirm participation in the research study:
  The investigators are looking for the highest dose of the combination of study drugs that can be administered safely without severe or unmanageable side effects in participants that have CD52 positive aggressive lymphoma. Not everyone who participates in this research study will receive the same dose of the study drug. The dose given will depend on the number of participants who have been enrolled in the study prior and how well the dose was tolerated.
  * Cyclophosphamide
  * Alemtuzumab
  Interventions: Drug: Cyclophosphamide; Drug: Alemtuzumab

INTERVENTIONS:
Drug: Cyclophosphamide — The chemotherapy drugs will be given in the hospital. During the first cycle of treatment, participants will stay in the hospital until their blood counts have recovered after treatment. During cycles 2 and 3, participants may go home after chemotherapy if they are doing well. The length of each cycle is 28 days
  - Via IV Day 3
  Other Names: Endoxan; Cytoxan; Lyophilized Cytoxan; Neosar; Revimmune; Procytox; Cycloblastin
Drug: Alemtuzumab — * The chemotherapy drugs will be given in the hospital. During the first cycle of treatment, participants will stay in the hospital until their blood counts have recovered after treatment. During cycles 2 and 3, participants may go home after chemotherapy if they are doing well. The length of each cycle is 28 days
  * Alemtuzumab will be administered as follows:
    * IV Day 1
    * IV Day 2
    * Target dose IV on Day 3 and 4
  Other Names: Campath

SUMMARY:
This research study is studying a combination of chemotherapy drugs as a possible treatment for aggressive lymphoma that has not responded to standard treatment.

The names of the study interventions involved in this study are:

* Cyclophosphamide
* Alemtuzumab

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational intervention and also tries to define the appropriate dose of the investigational intervention to use for further studies. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved alemtuzumab for aggressive lymphoma but it has been approved for other uses.

In this research study, the investigators are studying the combination of cyclophosphamide and alemtuzumab in participants with several types of aggressive lymphoma which are positive for a protein called CD52, the target of alemtuzumab. Studies in laboratory models of CD52 positive lymphoma showed the combination of cyclophosphamide and alemtuzumab was very effective. Cyclophosphamide causes a specific type of immune cell, called a macrophage, to attack lymphoma cells treated with alemtuzumab. Both drugs have been used in participants with lymphoma but have not been previously combined in this way. The investigators hope to identify the highest dose of the drugs that can be safely given together and to see if the combination if effective in treating these lymphomas.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed non-Hodgkin lymphoma and be considered ineligible for standard curative therapeutic options, including high dose chemotherapy with autologous stem cell rescue.
* Participants with the following subtypes of CD52 positive non-Hodgkin lymphoma (defined as ≥ 50% positive staining by immunohistochemical staining or flow cytometry by local lab) will be considered eligible:
* High-grade B-cell lymphoma, with MYC and BCL2 and/or BCL6 rearrangements (DHL)
* DLBCL or high-grade B-cell lymphoma NOS or B-cell lymphoma unclassifiable with features intermediate between Burkitt lymphoma and diffuse large B-cell lymphoma with MYC and BCL2 protein over-expression by immunohistochemical (IHC) staining as defined by MYC expression in ≥ 40% of cells and BCL2 positivity ≥ 50% (DOL)
* Transformed lymphoma with MYC rearrangement by FISH or over-expression by IHC, as above
* CD52 positive mature T-cell lymphoproliferative disorder
* There is no limit to the prior number of chemotherapy regimens. Patients with prior autologous or allogeneic stem cell transplantation, as well as prior therapy with cyclophosphamide or alemtuzumab, are eligible.
* Age ≥ 18 and ≤75
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Participants must have normal organ and marrow function as defined by peripheral blood values below:

  * leukocytes ≥1,000/mcL
  * absolute neutrophil count ≥500/mcL
  * platelets ≥25,000/mcL
  * total bilirubin ≤ 2 × institutional upper limit of normal (ULN) unless related to Gilbert's disease
  * AST(SGOT)/ALT(SGPT) ≤ 3 × institutional ULN
  * creatinine clearance < 1.5 x institutional ULN
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 1 weeks (4 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Participants who are receiving any other investigational agents for their lymphoma.
* Participants receiving corticosteroids within the past 1 week.
* Participants with known active CNS involvement by lymphoma should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to cyclophosphamide or alemtuzumab
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled hematuria related to bladder injury or psychiatric illness/social situations that could limit compliance with study requirements.
* Pregnant women are excluded from this study because cyclophosphamide and alemtuzumab at these doses have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued. Negative serum pregnancy test will be required for women of childbearing potential.
* HIV-positive participants on combination antiretroviral therapy are ineligible because of the increased risk of lethal infections when treated with marrow-suppressive therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-07-30 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
MTD of Cyclophosphamide and Alemtuzumab | 28 days
  maximum tolerated dose of the combination of cyclophosphamide and alemtuzumab

SECONDARY OUTCOMES:
Overall Response Rate | 12 Months
  Non-Hodgkin Lymphoma Response Criteria, which will be reported descriptively
Complete Response Rate | 12 Months
  Non-Hodgkin Lymphoma Response Criteria, which will be reported descriptively
Progression Free Survival | up to 5 years
  Progression-free will be estimated using the method of Kaplan and Meier.
Overall Survival | up to 5 years
  Overall survival will be estimated using the method of Kaplan and Meier.
Response Rate | 28 Days
  Assess response by PET/CT and in the bone marrow after one cycle of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ann LaCasce, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No